CLINICAL TRIAL: NCT00000448
Title: Naltrexone: Consummatory Behaviors in Alcoholic Women
Brief Title: Naltrexone Treatment for Alcoholic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAOMA10225; R01AA010225 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Alcoholism; Eating Disorder
MeSH Terms: conditions — Alcoholism; Feeding and Eating Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects were given an inert placebo for 2 days, followed by daily doses of matching placebo for a total of 12 weeks.
  Interventions: Drug: Placebo
- Naltrexone (Experimental): Subjects were prescribed 25 mg naltrexone for 2 days, followed by daily doses of 50 mg of naltrexone for a total of 12 weeks.
  Interventions: Drug: naltrexone

INTERVENTIONS:
Drug: naltrexone — Naltrexone is an opioid receptor antagonist used primarily in the management of alcohol dependence and opioid dependence.
  Other Names: Revia; Depade
  Arms: Naltrexone
Drug: Placebo — A placebo is a simulated or otherwise medically ineffectual treatment for a disease or other medical condition intended to deceive the recipient.
  Arms: Placebo

SUMMARY:
This study will assess naltrexone's effectiveness in treating alcoholism in women and provide information on its potential value in treating eating disorders common among alcoholic women. Alcoholic women with and without both eating disorders and depression will be randomly assigned to placebo or naltrexone treatment. Each group will receive behavioral therapy for 12 weeks, with followup 6 months after treatment.

DETAILED DESCRIPTION:
Background: Despite important gender differences in drinking patterns, physiological effects of alcohol, and co-occurring psychiatric conditions, relatively little is known about the efficacy of naltrexone for the treatment of alcohol dependence in women. This study investigated the safety and efficacy of naltrexone in combination with Cognitive Behavioral Coping Skills Therapy (CBCST) in a sample of alcohol-dependent women, some with comorbid eating pathology.

Methods: One hundred three women meeting DSM-IV criteria for alcohol dependence (29 with comorbid eating disturbances) were randomized to receive either naltrexone or placebo for 12 weeks in addition to weekly group CBCST.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence. Abstinent from alcohol for a period of at least 5 days.
* Able to read English and complete study evaluations.
* A stable residence and a telephone to ensure that subjects can be located during the study.

Exclusion Criteria:

* Meets criteria for dependence on another psychoactive substance besides alcohol or nicotine.
* Regular use of psychoactive drugs except antidepressants.
* Current use of disulfiram (Antabuse).
* Psychotic or otherwise severely psychiatrically disabled.
* Significant underlying medical conditions such as cerebral, renal, thyroid, or cardiac pathology.
* Abstinent longer than 30 days prior to admission to program.
* Hepatocellular disease or elevated bilirubin levels.
* Individuals with present history of opiate abuse or who require the use of opioid analgesics.
* Women who are pregnant, nursing, or not using a reliable method of birth control.
* Women who are significantly overweight or significantly underweight.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 1995-10; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Time to first day of drinking | 12 week treatment period
Time to first day of heavy drinking | 12 weeks
  Defined as consuming 4 or more drinks during the 12-week period

SECONDARY OUTCOMES:
Percentage of days abstinent | 12 weeks of treatment
Percentage of heavy drinking days | 12 weeks of treatment
Beck Depression Index | 12 weeks of treatment
  The Beck Depression Inventory (BDI, BDI-1A, BDI-II), created by Dr. Aaron T. Beck, is a 21-question multiple-choice self-report inventory. Higher total scores indicate more severe depressive symptoms. This was administered bi-weekly throughout the treatment period.
Obsessive Compulsive Drinking Scale (OCDS) | Baseline, Month 1, 2, 3
  The OCDS was developed to reflect obsessionality and compulsivity related to craving and drinking behavior.
Eating Disorder Examination (EDE) | baseline, month 1, 2, 3
  The Eating Disorder Examination Interview (EDE) devised by Cooper & Fairburn (1987) is a semi-structured interview conducted by a clinician in the assessment of an eating disorder. The questions concern the frequency in which the patient engages in behaviors indicative of an eating disorder over a 28 day period. The test is scored on a 7 point scale from 0-6. With a zero score indicating not having engaged in the questioned behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie S O'Malley, PhD, Principal Investigator — Yale University
Locations (1):
- Substance Abuse Treatment Unit, Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Result] O'Malley SS, Sinha R, Grilo CM, Capone C, Farren CK, McKee SA, Rounsaville BJ, Wu R. Naltrexone and cognitive behavioral coping skills therapy for the treatment of alcohol drinking and eating disorder features in alcohol-dependent women: a randomized controlled trial. Alcohol Clin Exp Res. 2007 Apr;31(4):625-34. doi: 10.1111/j.1530-0277.2007.00347.x. PMID 17374042
- See also: Published paper — http://onlinelibrary.wiley.com/doi/10.1111/j.1530-0277.2007.00347.x/abstract;jsessionid=18A7C01A7A320EC10B8553D84B4C4A1F.f02t03